CLINICAL TRIAL: NCT04328831
Title: A Phase 1a/1b Study Evaluating the Safety, Tolerability and Preliminary Efficacy of IBI322 in Subjects With Advanced Malignant Tumors
Brief Title: Safety and Efficacy of IBI322 in Chinese Subjects With Advanced Malignant Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI322A101
Record Dates: First submitted 2020-03-24; First posted 2020-03-31 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Advanced Malignancies
Keywords: Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI322 (Other): Single arm
  Interventions: Biological: IBI322

INTERVENTIONS:
Biological: IBI322 — Recombinant anti-human CD47/PD-L1 bispecific antibody injection

SUMMARY:
This is a phase I study evaluating the safety, tolerability and preliminary efficacy of IBI322 in cancer subjects who failed standard treatment.

DETAILED DESCRIPTION:
Phase 1a/Ib study will be conducted to evaluate the tolerability, safety, PK, PD, immunogenicity and preliminary antitumor activity of IBI322 in China. Phase 1a is dose escalation and plans to enroll approximately 38-60 subjects with advanced malignant solid tumors who failed the standard treatment. Phase Ib is dose expansion, and plans to enroll approximately 180 subjects with advanced malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically/cytologically confirmed, locally advanced unresectable or metastatic tumors.
2. At least one evaluable lesion.
3. Male or female subject above 18 years old, no more than 75 years old.
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) performance status 0 or 1.
5. Must have adequate organ function

Exclusion Criteria:

1. Previous exposure to any anti-CD47 monoclonal antibody, SIRPα antibody, or CD47/SIRPα recombinant protein.
2. Previous exposure to any anti-programmed death receptor 1 (PD-1) or anti-programmed death ligand 1 (PD-L1) /anti-programmed death ligand 2 (PD-L2) antibodies
3. Subjects participating in another interventional clinical study, except for: observational (non-interventional) clinical studies or survival follow-up phase of interventional studies.
4. Patients who are on anticoagulants and /or require concomitant aspirin or other nonsteroids anti-inflammatory medications. Patients with a history of a bleeding diathesis (von Willebrand disease, end stage liver disease, hemophilia, etc.)
5. Subjects who have a history of blood transfusion within 2 weeks prior to the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Number of DLT | 28 days
Number of treatment related AEs | 90 days post last dose
Number of patients with response | Last patient enrolled+24 weeks

SECONDARY OUTCOMES:
PK parameters: The area under the curve (AUC) | Up to 90 days post last dose
PK parameters: Maximum concentration (Cmax) | Up to 90 days post last dose
PK parameters: Time at which maximum concentration (Tmax) | Up to 90 days post last dose
PK parameters: The half-life (t1/2) | Up to 90 days post last dose
Positive rate of ADA and Nab | Up to 90 days post last dose
Positive rate of Circulating Immune Complex | Up to last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer hospital Chinese academy of Medical sciences, Beijing, China